CLINICAL TRIAL: NCT00731952
Title: Phase I Study of Induction Therapy With VELCADE and Vorinostat in Patients With Surgically Resectable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Benjamin Kozower, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12472
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: surgically resectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade and Vorinostat (Experimental): Subjects will receive one of 3 doses of Velcade (at a dose of 1.0 - 1.6 mg/m2 once weekly for 3 weeks) and one of 4 doses of Vorinostat (at a dose of 100mg every day 3 times a week for 3 weeks to 300mg twice per day, 3 times per week for 3 weeks). Doses determined by a predetermined escalation schedule.
  Interventions: Drug: Velcade and Vorinostat

INTERVENTIONS:
Drug: Velcade and Vorinostat — Subjects will receive one of 3 doses of Velcade (at a dose of 1.0 - 1.6 mg/m2 once weekly for 3 weeks) and one of 4 doses of Vorinostat (at a dose of 100mg every day 3 times a week for 3 weeks to 300mg twice per day, 3 times per week for 3 weeks). Doses determined by a predetermined escalation schedule.

SUMMARY:
The purpose of this study is to find out what effects (both good and bad) two medications (VELCADE and Vorinostat) have on patients who have certain types of lung cancer. The study is "dose escalating" meaning that patients will receive different doses of medication depending on when they enter the study. Participation in the study will last approximately 3 months and will include an initial screening visit, a visit once each week for 3 weeks to receive the study medications, and then 2 additional visits around the time of your surgery to remove your lung cancer tumor.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed NSCLC (clinical stage IB, IIA, IIB, IIIA, or selected IIIB (T4N0-1M0)), exclusive of patients with MPE
* Planned surgical resection
* Age > 18 years
* ECOG performance status 0-1
* Patient has adequate organ and marrow function, as defined below:
* Patient has a platelet count of > 100 x 109/L
* Patient has a WBC count of > 3.5 x 109/L
* Patient has an absolute neutrophil count of > 1.5 x 109/L
* Patient has hemoglobin of > 8 gm/dl. Patients may receive transfusions, erythropoietin or darbepoetin to achieve this hemoglobin level.
* Patient has a serum creatinine of < 2.0 mg/dL
* Patient has AST < 1.5 x ULN
* Patient has bilirubin < 1.5 x ULN
* Patient has INR < 1.5 x ULN
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria

* Previous chemotherapy or radiation therapy within 5 years before enrollment.
* Prior history of treatment for a known NSCLC within the last 5 years of if > 5 years but still thought by the investigator to represent recurrent disease.
* Prior exposure to either Velcade or Vorinostat
* Prior exposure to any HDAC inhibitors within the previous 30 days. Patients who have received such agents for other indications may enroll after 30-day wash-out period. Subject may not take any other HDAC inhibitor during this trial.
* Patient has >/= Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to VELCADE, boron or mannitol.
* Patient has known allergy to any component of Vorinostat (MK-0683)
* Female subject is pregnant or breast-feeding. Confirm by a negative serum B-hCG pregnancy test result obtained during screening (not required for post-menopausal or surgically sterilized women).
* Patient is participating or has participated in another investigational trial, and has received other investigational drugs/therapies within 30 days of enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has history of GI surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs.
* Subject is currently taking herbal remedy and/or homeopathic agent which cannot (or the patient is unwilling) be discontinued during the conduct of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-06; Primary Completion 2012-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | 30 days post surgical resection

SECONDARY OUTCOMES:
Tumor response | Day 22

CONTACTS AND LOCATIONS:
Overall Officials: David R Jones, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States